CLINICAL TRIAL: NCT05464628
Title: A Phase 1, Open-Label, Drug-Drug Interaction, Study to Evaluate the Effect of ASC42 on the Pharmacokinetics of Atorvastatin Tablets in Healthy Volunteers (HVs)
Brief Title: Drug Interaction Study of ASC42 With Atorvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gannex Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ASC42-103
Record Dates: First submitted 2022-07-12; First posted 2022-07-19 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: ASC42; Atorvastatin
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atorvastatin and ASC42 (Experimental): Atorvastatin followed by ASC42 daily followed by separate co-administration of atorvastatin.
  Interventions: Drug: Atorvastatin; Drug: ASC42

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin followed by ASC42 daily followed by separate co-administration of atorvastatin
  Other Names: Lipitor
Drug: ASC42 — Atorvastatin followed by ASC42 daily followed by separate co-administration of atorvastatin

SUMMARY:
The purpose of this study is to determine whether ASC42 alters the pharmacokinetics of atorvastatin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between 18 to 65 years of age
* Willing and able to give informed consent prior to any procedures
* Weight at least 50 kg and have a body mass index (BMI) within the range of 19-32 kg/m^2, inclusive at screening.
* A female participant is eligible to participate in this study if: She is of non-childbearing potential. She is of childbearing potential and is non-pregnant or non-lactating and willing to use adequate contraception from screening until 30 days after the End of Study visit.
* Physical examination and vital signs are within normal range or slightly abnormal but nonclinical significance.

Exclusion Criteria:

* Females with childbearing potential if no dual safe anticontraception method is provided.
* Male subjects whose female partner is currently pregnant or wanting to become pregnant or sexually active subjects if methods of contraception are not used during the trial and for 30 days following their final study drug.
* ALT or AST >ULN or Direct bilirubin >ULN
* Total Bilirubin >ULN with any single parameters of ALT, AST, ALP or GGT > ULN
* Elevated creatine kinase (CK) at screening (one repeat test allowed)
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or may jeopardize the safety of the participants.
* Platelet count <150,000/mcL or INR> 1.2
* History of , or current electrocardiogram abnormalities, arrythmias or heart valve diseases.
* History of drug or food allergies that caused severe hypersensitivity.
* History of intolerance to or adverse event reaction to a statin, or history of myopathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the pharmacokinetics (PK) of atorvastatin and its two metabolites by Peak Plasma Concentration (Cmax) in the presence or absence of ASC42 | 120 hours
Evaluate the pharmacokinetics (PK) of Atorvastatin and its two metabolites in the presence of ASC42 by Area under the curve from the time of dosing extrapolated to infinity (AUC(0-inf)) | 120 hours
Evaluate the pharmacokinetics (PK) of atorvastatin and its two metabolites by time to peak plasma concentration (Tmax) in the presence or absence of ASC42 | 120 hours

SECONDARY OUTCOMES:
Safety and tolerability of Atorvastatin in the presence of ASC42 evaluated by incidence of treatment emergent adverse events (TEAEs) | Baseline to Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, San Antonio, Texas, United States